CLINICAL TRIAL: NCT00002324
Title: A Multi-Center, Placebo-Controlled, Double-Blind, Randomized Trial Comparing the Activity, Safety, and Tolerance of 1) 400 Mg Nevirapine in Combination With 500-600 Mg Zidovudine Versus Zidovudine Alone in Asymptomatic HIV-1 Infected Patients With 3-24 Months of Prior Zidovudine Therapy and 200-500 CD4 Cells/mm3 and 2) 400 Mg Nevirapine Versus Nevirapine Placebo in Asymptomatic HIV-1 Nucleoside Naive Patients With 200-500 CD4 Cells/mm3
Brief Title: The Safety and Effectiveness of Nevirapine and Zidovudine, Given Separately and Together, in HIV-1 Infected Patients Who Have No Symptoms of the Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 200C; 1038
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-08

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; AIDS-Related Complex; Zidovudine; Nevirapine
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Nevirapine; Zidovudine

INTERVENTIONS:
Drug: Nevirapine
Drug: Zidovudine

SUMMARY:
PRIMARY: To compare the effect of nevirapine versus placebo alone or in combination with zidovudine (AZT) on CD4 T-cell count and percentage after 3 and 6 months of treatment. To evaluate the safety and tolerance of nevirapine alone or in combination with AZT.

SECONDARY: To compare the effects of the various treatment combinations on virologic and immunologic markers.

DETAILED DESCRIPTION:
In Part I, patients who have had prior AZT therapy receive either nevirapine or placebo in combination with AZT. In Part II, patients who are nucleoside naive receive either nevirapine or matching placebo. After 6 months, patients receive open-label nevirapine.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* PCP prophylaxis (trimethoprim-sulfamethoxazole, dapsone, or aerosolized pentamidine), at the discretion of the investigator.
* Antifungal prophylaxis with oral fluconazole or ketoconazole.
* Antiviral prophylaxis for herpes simplex virus with <= 1000 mg/day oral acyclovir.
* Dilantin for prevention and treatment of seizures.

Patients must have:

* Asymptomatic HIV-1 infection, with positive serum antibody to HIV-1 as determined by ELISA or Western blot.
* CD4 count 200-500 cells/mm3 within 4-28 days prior to study entry.
* No conditions indicative of AIDS.
* None of the constitutional symptoms that are specifically excluded.
* Prior AZT for 3-24 months (amended 04/04/94) immediately prior to study entry (Part I) OR no prior AZT (Part II).
* Consent of parent or guardian if less than 18 years of age.

NOTE:

* Co-enrollment in a protocol involving another investigational drug or biologic is not permitted.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Malignancy other than limited cutaneous basal cell carcinoma.
* Psychiatric condition sufficient to impair compliance with protocol requirements.

Concurrent Medication:

Excluded:

* Investigational drugs other than study drugs.
* Systemic glucocorticoids and steroid hormones.
* Dicumarol, warfarin, and other anticoagulant medications.
* Cimetidine.
* Tolbutamide.
* Doxycycline.
* Chloramphenicol.
* Phenobarbital and other barbiturates.
* Foscarnet.
* Erythromycin.
* Amoxicillin-clavulanate (Augmentin).
* Ticarcillin clavulanate (Timentin).
* Biologic response modifiers (alpha interferon, IL-2, immune modulators).

Patients with the following condition are excluded:

History of other clinically important disease (i.e., one that precludes participation in the study).

Prior Medication:

Excluded:

* Antiretroviral medications other than AZT.

Excluded within 4 weeks prior to study entry:

* Immunosuppressive or cytotoxic drugs or other experimental drugs.
* Systemic glucocorticoids and steroid hormones.
* Dicumarol, warfarin, and other anticoagulant medications.
* Cimetidine.
* Tolbutamide.
* Doxycycline.
* Chloramphenicol.
* Phenobarbital and other barbiturates.
* Foscarnet.
* Erythromycin.
* Amoxicillin-clavulanate (Augmentin).
* Ticarcillin clavulanate (Timentin).
* Biologic response modifiers (alpha interferon, IL-2, immune modulators).

Required (for patients in Part I):

* Prior AZT at 500-600 mg daily for at least 3 months but not more than 24 months immediately prior to study entry.

Chronic use of alcohol or drugs sufficient to impair compliance with protocol requirements.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - UCSD Treatment Ctr, San Diego, California
  - Saint Francis Mem Hosp, San Francisco, California
  - Wilmington Hosp, Wilmington, Delaware
  - Community Research Initiative of South Florida, Coral Gables, Florida
  - Goodgame Med Group, Maitland, Florida
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - Chandler Med Ctr, Lexington, Kentucky
  - Kansas City AIDS Research Consortium, Kansas City, Missouri
  - Community Research Initiative on AIDS, New York, New York
  - Med College of Ohio, Toledo, Ohio
  - Associates Med and Mental Health, Tulsa, Oklahoma
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Dr Alfred F Burnside Jr, Columbia, South Carolina
  - Nelson-Tebedo Community Clinic, Dallas, Texas
  - Houston Clinical Research Network, Houston, Texas
  - Univ of Utah School of Medicine, Salt Lake City, Utah
  - Infectious Disease Physicians Inc, Annandale, Virginia
  - Richmond AIDS Consortium, Richmond, Virginia

REFERENCES:
- [Background] Pollard R . Surrogate marker response to NVP/ZDV or ZDV in a blinded clinical trial: correlation to changes in HIV isolate phenotypic susceptibility to NVP and ZDV. Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:113